CLINICAL TRIAL: NCT04226612
Title: Association of Inpatient Blood Pressure Levels With In-hospital Adverse Events(APPLE Study)
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018570H(R1)
Record Dates: First submitted 2019-12-24; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; Inpatient; Adverse Events; All-cause mortality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate the association between inpatient blood pressure levels and in-hosopital adverse outcomes.

DETAILED DESCRIPTION:
Study population includes subjects who are hospitalized due to illness, of any race or ethnicity, any of age.The primary outcome is all-cause mortality occured in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with all age or race;
* Have blood pressure data.

Exclusion Criteria:

* Non-patients；
* Death outside the hospital；
* Missing blood pressure data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | during the procedure
  All-cause mortality was confirmed through a combination of hospital medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ying-qing, PhD, Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Feng Ying-qing, Guangzhou, Guangdong, China